CLINICAL TRIAL: NCT00743275
Title: Immunogenicity and Safety Among Adults of the Inactivated, Split-Virion Influenza Vaccine, Northern Hemisphere 2008-2009 Formulation (Intramuscular Route)
Brief Title: A Study to Evaluate the Safety and Immune Responses to Fluzone® Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GRC41
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants received one dose of Fluzone® vaccine on Day 0.
  Interventions: Biological: Split, Inactivated, Trivalent Influenza vaccine (Fluzone®)

INTERVENTIONS:
Biological: Split, Inactivated, Trivalent Influenza vaccine (Fluzone®) — 0.5 mL, intramuscular
  Other Names: Fluzone®

SUMMARY:
To describe the safety of the inactivated, split-virion influenza vaccine, 2008-2009 formulation.

To evaluate the compliance, in terms of immunogenicity, of the inactivated, split-virion influenza vaccine 2008-2009 formulation with the requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or older on the day of inclusion.
* Participant willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Participant in reasonably good health as assessed by the Investigator.
* Participant willing and able to give informed consent.
* For a woman, inability to bear a child or negative serum/urine pregnancy test.

Exclusion Criteria:

* Self-reported allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* An acute illness with or without fever in the 72 hours preceding enrollment in the trial.
* Clinically significant findings in vital signs (including temperature ≥ 99.5°F oral) or review of systems.
* Self-reported history of severe adverse event to any influenza vaccine.
* Laboratory-confirmed influenza infection or vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 2.
* Participation in any other interventional drug or vaccine trial within the 30 days preceding or during enrollment into this study.*
* Immunocompromising condition or immunosuppressive therapy (including systemic steroid use for 2 weeks or more), cancer chemotherapy, or radiation therapy at the time of enrollment, planned during the period of this study, or at any time within the past 6 months.
* Receipt of blood or blood products within the 3 months preceding enrollment in the study.
* Diabetes mellitus requiring pharmacological control.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing potential, a positive urine pregnancy test, breast feeding, or not using a medically approved and reliable form of contraception (oral contraceptives or double barrier method) for the duration of the trial.
* Current use of alcohol or recreational drugs that may interfere with the subject's ability to comply with trial procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Prior personal history of Guillain-Barré syndrome. * Subjects enrolled into this study will not be prohibited from donating blood for non-interventional studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 26 August to 03 September 2008 at one US clinical center.
Pre-assignment Details: A total of 122 participants who met the inclusion and exclusion criteria were enrolled. Of these, 120 participants were vaccinated.
Groups:
- Age 18-60 Years; Age 61 Years and Older: Participants received one dose of Fluzone® vaccine on Day 0.
Period: Overall Study
Arm/Group | Age 18-60 Years | Age 61 Years and Older
Started | 59 | 61
Completed | 59 | 60
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 18-60 Years | Age 61 Years and Older | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 8 | 67
  >=65 years | 0 | 53 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (12.14) | 74.7 (7.67) | 59.2 (18.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 14 | 23 | 37
Region of Enrollment [Number; unit: participants]
  United States | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Solicited Injection Site Solicited Systemic Reactions Post-vaccination With Fluzone® Vaccine.
Description: Solicited Injection Site Reaction: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited Systemic Reaction: Fever (temperature), Headache, Malaise, Myalgia, and Shivering
Time Frame: Days 0-3 post-vaccination
Population: Safety profile was assessed in the intent-to-treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | Age 18-60 Years | Age 61 Years and Older
Number analyzed (Participants) | 59 | 61
Participants
  Any Solicited Injection Site Reaction | 35 | 18
  Any Pain | 34 | 16
  Grade 3 Pain (Incapacitating) | 0 | 1
  Any Erythema (Redness) | 7 | 2
  Grade 3 Erythema (Redness) | 0 | 0
  Any Swelling | 4 | 1
  Grade 3 Swelling (≥ 5 cm) | 0 | 1
  Any Induration | 5 | 1
  Grade 3 Induration (≥ 5 cm) | 0 | 0
  Any Ecchymosis | 2 | 1
  Grade 3 Ecchymosis (≥ 5 cm) | 0 | 0
  Any Solicited Systemic Reaction | 25 | 14
  Any Fever | 1 | 0
  Grade 3 Fever (> 102.2 ºF) | 0 | 0
  Any Headache | 17 | 6
  Grade 3 Headache | 1 | 0
  Any Malaise | 9 | 2
  Grade 3 Malaise (Prevents daily activities) | 1 | 0
  Any Myalgia | 19 | 10
  Grade 3 Myalgia (Prevents daily activities) | 1 | 1
  Any Shivering | 4 | 0
  Grade 3 Shivering (Prevents daily activities) | 0 | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) for the 3 Influenza Strains Pre- and Post-vaccination With Fluzone® Vaccine 2008-2009 Formulation
Time Frame: Day 0 and 21 days post-vaccination
Population: Analysis of Geometric Mean Titers was in the per-protocol population. (Participants that did not provide both pre- and post- vaccination serum samples within the specified time window were excluded from analysis)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Age 18-60 Years | Age 61 Years and Older
Number analyzed (Participants) | 50 | 49
Titers
  A/Brisbane/59/2007 (H1N1) IVR-148 Pre-dose | 26.9 [18.8 to 38.6] | 16.9 [13.3 to 21.4]
  A/Uruguay (H3N2) X-175-C Pre-dose | 34.9 [22.5 to 54.2] | 31.5 [21.5 to 46.0]
  B/Florida/04/2006 Pre-dose | 28.5 [21.0 to 38.6] | 21.6 [16.6 to 28.1]
  A/Brisbane/59/2007 (H1N1) IVR-148 Post-dose | 130.9 [91.1 to 188.1] | 46.1 [35.0 to 60.7]
  A/Uruguay (H3N2) X-175-C Post-dose | 528.7 [351.1 to 796.3] | 300.3 [217.9 to 413.7]
  B/Florida/04/2006 Post-dose | 84.0 [64.9 to 108.6] | 56.2 [40.9 to 77.2]

3. Primary Outcome: Percentage of Participants With at Least 1:40 Hemagglutination Inhibition Antibody Titer Post-Vaccination With Fluzone® Vaccine (Seroprotection)
Description: Seroprotection was defined as post-vaccination titer value of ≥ 1:40.
Time Frame: 21 days post-vaccination
Population: Analysis of seroprotection was in the per-protocol population. (Participants that did not provide both pre- and post- vaccination serum samples within the specified time window were excluded from analysis)
Measure: Number; unit: Percentage of Participants
Arm/Group | Age 18-60 Years | Age 61 Years and Older
Number analyzed (Participants) | 50 | 49
Percentage of Participants
  A/Brisbane/59/2007 (H1N1) IVR-148 | 88 | 63
  A/Uruguay (H3N2) X-175-C | 98 | 98
  B/Florida/04/2006 | 82 | 67

4. Primary Outcome: Percentage of Participants With at Least a 4-Fold Rise in Hemagglutination Inhibition Antibody Titer Post-Vaccination With Fluzone Vaccine (Seroconversion)
Description: Seroconversion was defined as a four-fold rise in titers or greater from baseline. If the baseline titer value is < 10, then 10 is used as the baseline value for the purposes of this calculation
Time Frame: 21 days post-vaccination
Population: Analysis of seroconversion was in the per-protocol population. (Participants that did not provide both pre- and post- vaccination serum samples within the specified time window were excluded from analysis)
Measure: Number; unit: Percentage of Participants
Arm/Group | Age 18-60 Years | Age 61 Years and Older
Number analyzed (Participants) | 50 | 49
Percentage of Participants
  A/Brisbane/59/2007 (H1N1) IVR-148 | 42 | 33
  A/Uruguay (H3N2) X 175-C | 77 | 84
  B/Florida/04/2006 | 36 | 31

ADVERSE EVENTS:
Time Frame: Adverse events data were collected throughout the study from Day 0 to Day 21.
Arm/Group | Age 18-60 Years | Age 61 Years and Older
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 34/59 | 16/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 18-60 Years (N=59) | Age 61 Years and Older (N=61)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Injection site pain (General disorders) | 34 (34) | 16 (16)
Injection site erythema (General disorders) | 7 (7) | 2 (2)
Injection site swelling (General disorders) | 4 (4) | 1 (1)
Injection site induration (General disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 17 (17) | 6 (6)
Malaise (General disorders) | 9 (9) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 10 (10)
Chills (General disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications